CLINICAL TRIAL: NCT02766010
Title: A Comparative Clinical Study to Assess the Accuracy of TensorTip MTX, a Non Invasive Device for the Measurement of Physiological and Hematological Parameters
Brief Title: A Comparative Clinical Study to Assess the Accuracy of TensorTip MTX, a Non Invasive Device
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Cnoga Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CM-CL-P-PHY-002
Record Dates: First submitted 2016-03-28; First posted 2016-05-09 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2016-04

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group A TensorTip (Experimental): Male or female, age > 18
  Interventions: Device: TensorTip

INTERVENTIONS:
Device: TensorTip — Non Invasive screening of various physiological and hematological parameters.
  Other Names: Cnoga Medical Ltd. h SofTouch; SoftTouc

SUMMARY:
1. Aim- This study is aimed to access the accuracy of TensorTip MTX device measuring Hemoglobin A1C, Oxygen Concentration and Saturation ,Carbon Dioxide, Blood pH, Hemoglobin, Hematocrit, Red Cells Count, platelets, Blood Urea Nitrogen, Sodium, Potassium, Chloride, total bilirubin, cholesterol (HDL, LDL), Serum Creatinine, Peripheral Pulse Rate, Blood Pressure, Mean Arterial Pressure, cardiac output, cardiac index, stoke volume and blood gases compared with the simultaneous results from hospital references device (when available)
2. Hypothesis- Human physiological biomarkers may be measured from the color distribution of the internal or external (skin) tissue. The technology of the TensorTip device is based on the color distribution of the peripheral blood tissue, which enables the measurement of certain biomarkers and vital signs under consideration

DETAILED DESCRIPTION:
1. This is a comparative clinical trial in which the measurements obtained by the TensorTip device will be compared with those obtained by the reference devices used by the hospital on daily or periodic monitoring (the devices will be identified by name and version at the final report).
2. Eligible real time color signal obtained by the TensorTip during the measurement shall be recorded simultaneously with the measurements obtained by the reference devices (as described in the above point).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age > 18
2. Agree to sign voluntary inform consent.

Exclusion Criteria:

1. Refusal to sign an informed consent and to participate in the study.
2. Below the age of 18.
3. Finger size not suitable for the measurement chamber.
4. Injured skin in the measurement site.
5. Long fingernails

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-05-22 (Actual); Primary Completion 2016-08-29 (Actual); Study Completion 2016-08-29 (Actual)

PRIMARY OUTCOMES:
blood pressure measurement of the TensorTip against hospital readings | 3 months

IPD SHARING:
Plan to Share IPD: Undecided